CLINICAL TRIAL: NCT05752331
Title: Feasibility of Personalised Health Behaviour Coaching to Support Symptoms and Activities of Daily Living in Those With Long COVID-19.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCACORN
Record Dates: First submitted 2023-02-28; First posted 2023-03-02 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Long COVID
Keywords: Physical activity; Fatigue; Breathlessness
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity; Fatigue; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity behavioural modification (Experimental): The 8-week PA behavioural modification intervention will focus on engaging participants in ADL and lowering sedentary time. Each participant will receive one semi-structured motivational interview at baseline to discuss favourite activities and barriers and facilitators to PA. Participants will produce an individualised action plan following the interview that will be followed throughout the intervention to allow an individualised approach to take place. Participants will then be provided with a low-cost pedometer and PA diary to self-monitor and record daily PA. The PA diary will provide examples of various activities that can be done in and around the house, with an emphasis placed on simple, effective movements to reduce sedentary time. Following this, a researcher will conduct weekly virtual meetings with the participant to discuss the past weeks PA levels and provide future individualised goals to promote ADL.
  Interventions: Behavioral: Physical activity behavioural modification
- Usual Care (No Intervention): All participants will be notified of the government 'your Covid recovery' programme (usual care) which provides details and support on managing long term symptoms of Covid-19.

INTERVENTIONS:
Behavioral: Physical activity behavioural modification — 8-week intervention consisting motivational interview, individualised action plan and weekly consultations regarding activities of daily living and symptom management.
  Arms: Physical activity behavioural modification

SUMMARY:
This pilot RCT aims to assess whether a simple PA behavioural modification intervention can be delivered safely and feasibly to individuals with Long COVID suffering long standing symptoms with concerns regarding their ability to perform activities of daily living.

Participants will be randomised to receive an 8-week physical activity behavioural modification intervention alongside usual care or usual care alone. The primary outcome for this study is to assess the safety and feasibility of the intervention, including recruitment targets, randomisation, completion rates and acceptability to the study.

DETAILED DESCRIPTION:
Coronavirus (COVID-19) is an infectious disease caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), infecting over 254 million people worldwide to date. While the majority of positive cases have uncomplicated recoveries, some have prolonged periods of persistent symptoms, referred to as Long Covid (symptoms ≥12 weeks). Many of the typical symptoms observed in those with Long Covid (fatigue, shortness of breath & cognitive dysfunction) are compounded by deconditioning associated with a sedentary lifestyle. This has become a major concern due to enforced lockdowns impacting individuals' abilities to conduct activities of daily living (ADL), causing many to resort to sedentary lifestyles. Worryingly, a significant association between sedentary behaviour and mental wellbeing has been highlighted in those with Long Covid, negatively impacting both physical and psychological symptoms.

Current research has focused on the lived experiences of people with Long Covid and how they undertake ADL. Key barriers to ADL included an ever-increasing depletion of energy reserves during low intensity physical activity (PA), an inability to manage symptoms of fatigue and breathlessness, and high levels of anxiety associated with safely pursing the potential benefits of PA. What's promising is that after expressing these barriers many individuals wished to prioritise recovery and return to a greater level of ADL as it provided a sense of normalisation and boosted overall mood. Subsequently, future research needs to investigate potential interventions which positively impact upon the sedentary behaviour of those with Long Covid and increase their ability to conduct ADL. Importantly, interventions of this nature must focus on reducing the symptoms of Long Covid during PA in order to promote a sense of safety while individuals purse the benefits of PA.

Therefore, this pilot randomised control trial (RCT) aims to assess whether a simple PA behavioural modification intervention can be delivered safely and feasibly to individuals with Long Covid who haven't been hospitalised due to Covid-19.

This pilot RCT will constitute a two parallel group study, with individuals randomised 1:1 to either an 8-week PA behavioural modification intervention alongside usual care (intervention group) or usual care alone (control group). Individuals with long standing symptoms (≥12 weeks) of COVID-19 who haven't previously been hospitalised will be recruited through university (staff & students) and community based non-NHS groups in order to avoid lengthy NHS ethical approval during feasibility. Eligible participants will attend 2 visits to a BU laboratory at baseline (week 0) and study completion (week 9) to complete all physiological and psychological measures (detailed below).

The 8-week PA behavioural modification intervention will focus on engaging participants in ADL and lowering sedentary time. Each participant will receive one semi-structured motivational interview at baseline to discuss favourite activities and barriers and facilitators to PA. Participants will produce an individualised action plan following the interview that will be followed throughout the intervention to allow an individualised approach to take place. Participants will then be provided with a low-cost pedometer and PA diary to self-monitor and record daily PA. The PA diary will provide examples of various activities that can be done in and around the house, with an emphasis placed on simple, effective movements to reduce sedentary time. Following this, a researcher will conduct weekly virtual meetings with the participant to discuss the past weeks PA levels and provide future individualised goals to promote ADL. All participants will be notified of the government 'your Covid recovery' programme (usual care) which provides details and support on managing long term symptoms of Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* People who are aged 18 years or older
* Have experienced at least one long COVID symptom for 12 weeks or longer
* Additionally meet at least one of the following criteria: 1) positive SARS-CoV-2 PCR or antigen test (positive COVID-19 test) during the acute phase of illness; 2) positive SARS-CoV-2 antibody test at any time point; 3) symptoms consistent with SARS-CoV-2 (COVID-19) infection during the acute phase.

Exclusion Criteria:

* Individuals who have previously been admitted to an intensive care unit (ICU) due to SARS-CoV-2
* Receiving palliative or end-of-life care
* Are actively participating in another research trial focused on long COVID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Participant recruitment | 8 weeks
  At least 40% of eligible participants recruited to the study
Participant randomisation | 8 weeks
  At least 80% of participants randomised following informed consent
Participant completion | 8 weeks
  At least 80% of randomised participants completing the intervention period and post assessment visit
Participant acceptability | 8 weeks
  Assessed through a project tailored questionnaire on completing of the study

SECONDARY OUTCOMES:
Objective physical activity | 8-weeks
  Accelerometer steps/day, Movement intensity & time spend in domains of activity.
Exercise capacity | 8-weeks
  Incremental shuttle walk test
Muscular strength and endurance | 8-weeks
  30-second sit to stand test and hand grip dynamometry
Lung Function | 8-weeks
  Spirometry measures of FEV1 and FVC
Health related quality of life | 8-weeks
  EQ-5D-5L
Breathlessness | 8-weeks
  COPD Assessment Test (CAT) and MRC dyspnea scale
Fatigue | 8 weeks
  Chalder fatigue scale
Anxiety and Depression | 8-weeks
  Hospital anxiety and depression scale
Cognitive impairment | 8-weeks
  MoCA

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Armstrong, Principal Investigator — Bournemouth University
Locations (1):
- Bournemouth University, Bournemouth, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: No